CLINICAL TRIAL: NCT03037450
Title: Miniinvasive Corneal Neurotization. A Pilot Study.
Acronym: MICORNE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The reasons for stopping the research are :
  * Inclusion difficulties (demanding inclusion and exclusion criteria),
  * The Covid-19 pandemic
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6528
Record Dates: First submitted 2017-01-17; First posted 2017-01-31 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Neurotrophic Keratitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Miniinvasive corneal neurotization (Other)
  Interventions: Procedure: Miniinvasive corneal neurotization

INTERVENTIONS:
Procedure: Miniinvasive corneal neurotization — Neurotization of a neurotrophic cornea

SUMMARY:
Neurotrophic keratitis (NK) is a degenerative disease of the cornea due to the impairment of the nasociliary branch of the ophthalmic nerve. Reduced corneal sensation lead to several corneal lesions including spontaneous ulcerations, delayed wound healing, corneal scarring, neovascularization, thinning, perforation or infection. An important and permanent visual loss of is frequently associated with the condition. NK can be congenital or acquired. Its acquired forms can be due to traumatic, infectious (herpes, zoster), neoplastic or iatrogenic causes. There is currently no specific medical treatment. Surgical reconstruction techniques of sensory neurotizations have recently been described in young patients suffering traumatic, congenital or neoplastic NK using supratrochlear nerves as the sensory donor nerves and sural nerve as healthy graft. A neurotization involves the transfer of a healthy donor nerve segment into a tissue to reestablish either motor or sensory innervation. The aim of the present study is to assess the outcomes of a novel sensory neurotization technique for the treatment of severe NK in adult patients (Stages 2 and 3 of Mackie classification). Corneal neurotizations will be performed using either ipsilateral supraorbital nerve as donor nerve (direct neurotization) or contralateral supraorbital nerve as donor nerve and a segment of the lateral antebrachial cutaneous nerve as graft. Small-size skin incisions (less than 3 centimeters) will be made in one or both eyebrow and an endoscopic device will help the surgeons to localize and dissect the supraorbital nerve. Donor nerves or graft will be sutured to the neurotrophic corneas. Adult patients with unilateral NK due to infectious, traumatic or iatrogenic causes will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18.
* NK stages 2 and 3 (Mackie's classification).
* Non-response to maximal medical treatment (lachrymal substitution, autologous serum).
* Postherpetic or post-zoster NK (Group 1).
* Postoperative NK (neurosurgery and trigeminal thermocoagulation) (Group 2).
* Posttraumatic NK (orbital trauma, ocular burn) (Group 3).
* No ocular hypertony in both eyes.
* Visual acuity > 20/40 on the contralateral eye.
* Written consent of the patient.
* Patient benefiting from national health coverage (either as a direct user or beneficiary).

Exclusion Criteria:

* Impossibility of general anesthesia.
* Herpetic or zoster recurrence in the 6 months prior surgery.
* Length of NK evolution > 5 years.
* Congenital NK.
* Bilateral NK.
* Other causes of NK: diabeta mellitus, amylosis, sarcoidosis, multiple sclerosis, vitamin A or B12 deficiency, Sjögren syndrome, GVH disease, topical NSAID, topical beta-blockers, history of refractive surgery.
* Mental illness.
* Adult with legal guardian or guardianship.
* Pregnancy.
* Breast-feeding.
* Patient's unable to understand informations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
Corneal sensation scores. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No